CLINICAL TRIAL: NCT02336334
Title: Measurement and Logging of Posturing Adherence of Patients After Intraocular Surgery With Gasendotamponades Using a Sensorsystem With Different Feedback-Methods
Brief Title: Evaluation of Posturing-Adherence in Patients After Intraocular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PosturingSensor
Record Dates: First submitted 2014-12-08; First posted 2015-01-13 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Retina; Lesion; Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With macular hole (Experimental): Inclusion of patients with macular holes and randomized allocation to sensor-types and information-types
  Interventions:
  Positioning measurement Patient feedback Usefulness of a sketch Closure rate of macular holes
  Interventions: Device: Positioning measurement; Device: Patient feedback; Procedure: Usefulness of a sketch; Device: Closure rate of macular holes
- Without macular hole (Experimental): Inclusion of patients without macular holes and randomized allocation to sensor-types and information-types
  Interventions:
  Positioning measurement Patient feedback Usefulness of a sketch
  Interventions: Device: Positioning measurement; Device: Patient feedback; Procedure: Usefulness of a sketch

INTERVENTIONS:
Device: Positioning measurement — Logging of posturing informations
Device: Patient feedback — Evaluation of patients questionary
Procedure: Usefulness of a sketch — Helping the patients to understand posturing positions by randomized allocation of sketches
Device: Closure rate of macular holes — closure rates of macular holes in the group with macular holes. Measurement using SD-OCT (spectral domain optical coherence tomography=
  Arms: With macular hole

SUMMARY:
Measuring and logging head positions of patients which underwent surgery with gasendotamponades.

DETAILED DESCRIPTION:
After surgery with gasendotamponades various positions are recommended to support the success of surgery. In patients with macular holes face-down-position is recommended. In patients with retinal detachment the recommended position depends on the region of the detachment.

The adherence of patients to follow this posturing instructions is very inhomogenous. Therefore the investigators want to measure the posturing by the use of a position-sensor. In some study arms the patients also receive a feedback from the sensor (tone, vibration) to correct the position.

The sensor-device was developed by the study-staff and is not commercial available. In addition there is no trade name. The patients safety of the used device was approved by the in house technical department.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* full thickness macular hole or retinal detachment
* informed consent

Exclusion Criteria:

* intraoperative complications with the need of other endotamponades
* combined treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2016-04 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Effective time of ideal posturing with different sensors-systems | up to 12 month
  Time (measured in minutes and in percent of 24h) with correct posturing in relation to the used sensor-type (with and without feedback)

SECONDARY OUTCOMES:
Time analysis with optimal posturing after detailed explanation of posturing positions | up to 12 month
  Time (measured in minutes and in percent of 24h) with correct posturing in patients which received an detailed posturing explanation (with graphics)
Analysis of time with optimal posturing for both Sensor-Feedback-Systems | up to 12 month
  Time (measured in minutes and in percent of 24h) with correct posturing depending on the used sensor-type (noise vs. vibration)
Closure rate of macular holes after 3 month as measured by optical coherence tomography (hole closed: yes or no) | up to 12 month
  Status of macular holes after 3 month in macular hole group measured by optical coherence tomography (hole closed: yes or no) and in relation to time with optimal posturing
Tolerability of sensor-systems for patients as measured by questionnaire | up to 12 month
  Using a questionnaire patients are asked to give their view on the tolerability of the used system.

CONTACTS AND LOCATIONS:
Locations (1):
- University Eye Hospital, Tübingen, Baden-Wurttemberg, Germany